CLINICAL TRIAL: NCT07102641
Title: PACESS: Post-cesarean Analgesia: Comparing Effectiveness of Staggered v. Simultaneous Therapies
Brief Title: Post-cesarean Analgesia: Comparing Effectiveness of Staggered v. Simultaneous Therapies
Acronym: PACESS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Whitney Bender, Assistant Professor, Department of Obstetrics and Gynecology, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2024-1669
Record Dates: First submitted 2025-07-25; First posted 2025-08-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Delivery; Postpartum Comfort; Postpartum Pain; Post-operative Pain; NSAIDs; Acetaminophen (D000082)
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Ketorolac; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Staggered (Active Comparator): Medications administered 3H apart (Staggered)
  Interventions: Drug: Acetaminophen; Drug: NSAID (Ketorolac/Ibuprofen)
- Simultaneous (Active Comparator): Medications administered at the same time. (Simultaneous)
  Interventions: Drug: Acetaminophen; Drug: NSAID (Ketorolac/Ibuprofen)

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 1000 mg q6H
Drug: NSAID (Ketorolac/Ibuprofen) — NSAID (ketorolac 30 mg q6H for first 24 hours post-op followed by ibuprofen 600 mg q6H)

SUMMARY:
Cesarean delivery is a commonly performed surgical procedure associated with worse postpartum pain when compared to vaginal birth. Uncontrolled postpartum pain is associated with increased neonatal and maternal risks. Multimodal non-opioid pain medications, including acetaminophen and non-steroidal anti-inflammatory drugs (NSAIDs) are the preferred first-line therapies. There is no standard practice, however, on best dosing schedules (ie staggered or different time v. simultaneous or same time). This protocol describes a randomized clinical trial aimed to determine whether staggered dosing of acetaminophen and NSAIDs in superior to simultaneous dosing in controlling post-cesarean pain.

DETAILED DESCRIPTION:
Cesarean delivery is a commonly performed surgical procedure. The rate of cesarean delivery (CD) is increasing in the US; cesarean accounted for 32% of all births in 2022. Parents who deliver via CD experience more pain than those who have a vaginal birth. Uncontrolled postpartum pain can be associated with an increased risk of physical complications including venous thrombosis, atelectasis, pneumonia as well as increased psychological distress. Poor postpartum pain control can also hinder infant-parental bonding and impact breastfeeding initiation or continuation.

Multiple strategies for post-operative pain management exist including opioid and non-opioid medications. Multimodal non-opioid medications are preferred as first-line therapies due to the short- and long-term risks associated with opioid pain medication. Acetaminophen and ibuprofen are most commonly utilized in the US. A meta-analysis of 21 studies enrolling 1909 post-operative patients examined the efficacy of NSAIDs and parecetamol in combination compared to each drug alone and found a significant reduction in pain intensity for combination therapy compared to each drug alone.

Both acetaminophen and ibuprofen can be given every 6 hours. Practices differ, however, on administering these medications at the same time or in a staggered fashion. To date, there are no trials comparing these different dosing schedules for post-cesarean delivery pain control.

ELIGIBILITY:
Inclusion Criteria:

* >/= 34 weeks gestation
* Singleton pregnancy
* Delivery via cesarean section under regional anesthesia

Exclusion Criteria:

* Contraindication to acetaminophen or NSAIDs
* Current or history of opioid use or misuse
* Intrauterine fetal demise
* Major congenital anomaly
* Conversion to general anesthesia intra-op or planned general anesthesia
* Mid-line vertical skin incision
* Receipt of intraoperative local analgesia such as Transversus Abdominis Plan (TAP) block or wound infiltration

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 825 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Postpartum pain control | 48 (+/- 2) hours postpartum
  Visual analog pain score (VAS) with movement. Scale ranges from 0-10 with 0 indicating no pain and 10 indicating worst possible pain
Opioid consumption | Postpartum Admission (From time of surgery to hospital discharge; typically 2-5 days)
  Opioid consumption (in total morphine milligram equivalents (MME))

SECONDARY OUTCOMES:
Postpartum pain at 6 hours | 6 hours (+/- 1 hour) post-op
  Visual analog pain score with rest. Scale ranges from 0-10 with 0 indicating no pain and 10 indicating worst possible pain
Postpartum pain at 12 hours | 12 hours (+/-2 hours) post-op
  Visual analog pain score with rest and movement. Scale ranges from 0-10 with 0 indicating no pain and 10 indicating worst possible pain
Postpartum pain at 24 hours | 24 hours (+/-2 hours) post-op
  Visual analog pain score with rest and movement. Scale ranges from 0-10 with 0 indicating no pain and 10 indicating worst possible pain
Postpartum pain at 48 hours | 48 hours (+/- 2 hours) post-op.
  Visual analog pain score with rest. Scale ranges from 0-10 with 0 indicating no pain and 10 indicating worst possible pain
Adequate pain control | by 48 hours (+/-2 hours) post-op
  Adequate pain control (Visual analog score <4). Scale ranges from 0-10 with 0 indicating no pain and 10 indicating worst possible pain
Length of stay | Admission to discharge (Typically 2-7 days)
  Duration of hospitalization
Infant feeding | At time of hospital discharge (Typically 1- 5 days post-op)
  Exclusive breastfeeding, combination feeding, or formula feeding
Patient satisfaction | Post-operative day #2-5.
  Patient satisfaction with pain control. Assessed via International Pain Outcomes (IPO) questionnaire. Scores for individual items in this questionnaire range from 0-10, with 0 indicating no symptoms and 10 indicating worst possible symptoms, OR from 0-100% for questions inquiring about time (0% being no time and 100% being all the time).
Opioid Prescription | At hospital discharge (Post-operative day #2-5)
  Need for opioid prescription (Yes or No) and amount (MME)
Home opioid | Post-operative day #10-14
  Home opioid use in the first week postpartum (Assessed by telephone call)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No